CLINICAL TRIAL: NCT05126446
Title: The Aorta Arch Stent Graft System Combined With the Endovascular Needle System in Situ Fenestration Technology in the Treatment of Aortic Dissection Involving the Aortic Arch
Brief Title: the Aorta Arch Stent Graft System Combined With the Endovascular Needle System in Situ Fenestration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTP86-01
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Aortic Dissection
Keywords: in situ fenestration; aortic dissection; aortic dissection involving the aortic arch
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- aortic dissection involving the aortic arch (Experimental): Aortic dissection involving the aortic arch was diagnosed in patients requiring revascularization of the aortic arch and its branches
  Interventions: Device: the Aorta Arch Stent Graft System combined with the Endovascular Needle System

INTERVENTIONS:
Device: the Aorta Arch Stent Graft System combined with the Endovascular Needle System — Patients who meet all the inclusion criteria and don't meet the exclusion criteria will be implanted with device

SUMMARY:
A prospective, multi-center, single-group target value method to evaluate the safety and effectiveness of the Aorta Arch Stent Graft System combined with the Endovascular Needle System in situ fenestration technology in the treatment of aortic dissection involving the aortic arch

DETAILED DESCRIPTION:
1. Clinical trials using prospective, multi-center, single-group target value design;
2. 120 subjects with aortic dissection requiring partial arch reconstruction will be enrolled in more than 30 centers in China, and they will meet the test enrollment requirements.
3. CTA examination was performed at baseline, 30 days, 6 months, 12 months, 36 months, and 60 months after surgery to determine the pathological status and the status of postoperative aortic and branch revascularization

ELIGIBILITY:
Inclusion criteria (to be selected if all of the following criteria are met)：

* 18 years old ≤age≤80 years old, no gender limitation;
* Diagnosis of aortic dissection and reconstruction of the left subclavian artery;
* The main branches and branches of the aortic arch at the lesion site have sufficient anatomical basis:

  * The diameter range of the near-end anchoring zone of the main body of the fixed mechanism: 21-46mm;
  * The length of the anchor zone near the principal part of the tunnel is ≥10mm;
  * The length of the anchor zone of the branching vessel of the convex target is ≥15mm;
  * The diameter range of the distal anchoring zone of the target branching vessel is 5-18mm.
* The patient has adequate surgical access vessels;
* Patients who understand the purpose of the study, voluntarily participate in and sign informed consent, and are willing to follow up.

Exclusion Criteria (If one of the following criteria is met, it will not be selected)：

* The patient is pregnant or breastfeeding;
* The patient had a history of cardiac surgery (congenital heart disease surgery, heart valve surgery, coronary heart disease surgery, thoracic aortic surgery, etc.), which would affect the implementation of this TEVAR surgery;
* The patient has been implanted or planned to be implanted with left ventricular auxiliary pump, interventional valve and other instruments, or is planning to undergo coronary intervention surgery, and aortic dissection is expected to affect the function of such instruments or such instruments will affect the operation of aortic dissection;
* Patients with severe hematoma on the aortic wall in the proximal anchoring area of the stent;
* Marfan syndrome and other connective tissue diseases, arteritis;
* Patients with a history of allergy to contrast agents, anesthetics, antiplatelet drugs, anticoagulants, nickel peptide alloys, and polytetrafluoroethylene materials;
* Patients with a history of cerebral infarction or myocardial infarction within 3 months before surgery;
* Patients with active bleeding and coagulopathy;
* Abnormal renal function: patients with preoperative creatinine > 2.5 times the normal upper limit value;
* Abnormal liver function: patients with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the normal upper limit value, or patients with serum total bilirubin (STB) > 2 times the normal upper limit value;
* Patients with end-stage diseases with a life expectancy of less than one year;
* patients with poor compliance considered by the investigator;
* Patients participating in other clinical trials at the same time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-25 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Primary safety end point of the Aorta Arch Stent Graft System: no Major Adverse events（MAE） occurrence within 30 days after surgery | Within 30 days after procedure
  MAE was defined as death related to aortic dissection, ischemic stroke, and paraplegia within 30 days after surgery
Primary efficacy endpoint of the Aorta Arch Stent Graft System: treatment success at 12 months after surgery | 12 months after procedure
  On the basis of successful surgery, the main and branch stents were unobstructed 12 months after surgery, with no internal leakage requiring intervention, no stent displacement (displacement ≤10mm), no new device-related rupture, and no device-induced aortic arch re-operation
Primary endpoint of the Endovascular Needle System: Immediate surgical success rate of the Endovascular Needle System | intraoperative
  Intraoperative DSA, the membrane was successfully broken in situ with the membrane rupture system, and the membrane rupture system was successfully withdrawn

CONTACTS AND LOCATIONS:
Overall Officials: Chang Shu, Professor, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- Xiangya Second Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Derived] Tan Y, Chen W, Li Z, Xu H, Zhao Y, Zhou D, Bai Y, Wang X, Xu T, Zhang Y, Xu J, Shu X. Early Results of a Single-Center Prospective Clinical Trial: In Situ Fenestration System for Aortic Dissection. Vasc Endovascular Surg. 2025 Aug;59(6):600-609. doi: 10.1177/15385744251330013. Epub 2025 Apr 27. PMID 40289333